CLINICAL TRIAL: NCT07100678
Title: Comparison Of Pretreatment Expectations and Posttreatment Satisfaction In Patients Receiving Porcelain-Fused-to-Metal Fixed Dental Prosthesis: A Quasi-Experimental Study
Brief Title: This Study Will Assess Whether the Treatment Provided by Dentist is Successful in Meeting the Expectations of Patient by Asking Questions Related to Aesthetics, Chewing Ability, Comfort and Phonetics Before and After Providing Treatment and the Patient Will Tell Through Visual Analog Scale
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber College of dentistry (Other)
Responsible Party: Principal Investigator, Zainab Rehman, Postgraduate Resident Prosthodontics, Khyber College of dentistry
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 46/RRB/KCD; Self, part of our training (Other: KCD)
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Patient Satisfaction
Keywords: patient satisfaction PFM Prosthodontics
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: This is a single-group, quasi-experimental study in which all participants will receive porcelain-fused-to-metal fixed dental prostheses. Pretreatment expectations and posttreatment satisfaction will be assessed within the same group to evaluate changes over time. No control or comparison group is included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Porcelain-Fused-to-Metal Fixed Dental Prosthesis (Experimental)
  Interventions: Procedure: Porcelain-Fused-to-Metal Fixed Dental Prosthesis

INTERVENTIONS:
Procedure: Porcelain-Fused-to-Metal Fixed Dental Prosthesis — This prosthesis consists of a metal substructure for strength and a porcelain coating for improved aesthetics. The treatment will be planned and delivered by prosthodontic specialist. The intervention is non-surgical

SUMMARY:
This study aims to assess patient satisfaction after receiving porcelain-fused-to-metal fixed dental prostheses. Patients will be asked about their expectations before treatment and their satisfaction afterward. The findings will help evaluate whether the treatment meets patient needs and guide improvements in dental care.

DETAILED DESCRIPTION:
This quasi-experimental study is designed to compare pretreatment expectations and posttreatment satisfaction in patients receiving porcelain-fused-to-metal fixed dental prostheses. The study will be conducted at the Prosthodontic Department of Khyber College of Dentistry, Peshawar, over a duration of six months.

A total of 120 partially edentulous patients aged 18 to 60 years, with no prior experience of fixed dental prostheses, will be included using a consecutive non-probability sampling technique. Prior to treatment, participants will be evaluated for their expectations regarding aesthetics, chewing ability, comfort, and phonetics using a validated questionnaire and a Visual Analogue Scale (VAS). Posttreatment satisfaction will be assessed using the same scale-on the day of prosthesis placement for aesthetics and phonetics, and after one week for chewing ability and comfort.

The aim is to evaluate whether there is a significant difference between what patients expect before treatment and how satisfied they are after receiving the prosthesis. The results will also help determine whether factors such as gender or age group influence satisfaction levels. This study seeks to contribute to more patient-centered treatment planning and improved outcomes in prosthodontic care.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous subjects between age group of 18 to 60 years.
* Patients who require and are willing to receive a fixed dental prosthesis.
* Patients with no experience of Fixed dental prosthesis previously.

Exclusion Criteria:

* Patients diagnosed with any psychological disorders (diagnosed by physician).
* Patients with facial anomalies like cleft lip and palate.
* Patients with skeletal class 2 or class 3.
* Patients with facial paralysis, stroke, and speech disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Patient Satisfaction Before and After Fixed Prosthodontic Treatment | Baseline (before prosthesis placement) and one week after prosthesis delivery.
  Patient satisfaction will be assessed in four domains-esthetics, comfort, chewing ability, and phonetics using a 10-point Visual Analogue Scale (VAS). Scores before treatment (expectation) and after treatment (satisfaction) will be compared to determine the change. . Each domain will be scored on a scale from 1 to 10, where 1 represents the lowest level of outcome and 10 represents the highest. The investigator will assess the results by adding all the marked values by the participant on VAS. Minimum and maximum values will be calculated from mean of scores on the basis of data collection results.

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Rehman, Postgraduate Resident(prostho), Principal Investigator — Khyber College of dentistry
Locations (1):
- Khyber College of Dentistry, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to privacy and confidentiality concerns, as well as institutional policies that restrict the dissemination of identifiable health information of study participants.

REFERENCES:
- [Background] Alqutaibi AY, Alharbi AF, Alharbi AM, Karbouji GA, Dagharire EY, Aboalrejal A. Pretreatment expectations and posttreatment satisfaction with different prosthodontic treatments in a Saudi population. Saudi J Oral Sci. 2022;9(1):63-71. DOI: 10.4103/sjoralsci.sjoralsci_52_21.
- See also: Pretreatment Expectations and Posttreatment Satisfaction with Different Prosthodontic Treatments in a Saudi Population — https://journals.lww.com/sjed/fulltext/2022/09010/pretreatment_expectations_and_posttreatment.11.aspx